CLINICAL TRIAL: NCT04790175
Title: Samsca Post-marketing General Drug Use-results Survey in Patients with Hyponatremia in Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH) in Japan
Brief Title: Samsca Post-marketing General Drug Use-results Survey in Patients with Hyponatremia in SIADH
Status: Recruiting | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-101-00348
Record Dates: First submitted 2021-02-25; First posted 2021-03-10 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Antidiuretic Hormone, Inappropriate Secretion
MeSH Terms: conditions — Inappropriate ADH Syndrome | interventions — Tolvaptan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tolvaptan (SAMSCA) — The usual adult dose of SAMSCA is 7.5 mg of tolvaptan once daily administered orally, increased stepwise to 60 mg daily until a desirable level of serum sodium concentration is achieved.

SUMMARY:
The purpose of this study is to confirm the safety of tolvaptan in patients with hyponatremia in syndrome of inappropriate antidiuretic hormone secretion (SIADH) in Japan

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a definite diagnosis of SIADH in reference to "Diagnostic and Treatment Manual of the Hypersecretion of Vasopressin (SIADH), Revised in 2018"

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Japan with hyponatremia in SIADH who are planned to be newly started on Samsca therapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Safety Information (Adverse Event) | 90 days from the initiation of tolvaptan treatment
  Any untoward medicinal occurrence in a patient or clinical study subject administered a Medicinal Product and which does not necessarily have a causal relationship with this treatment (ICH-E2A Guideline).
  An Adverse Event can therefore be any unfavorable and unintended sign (e.g. abnormal laboratory finding), symptom, or disease temporally associated with the use of a Medicinal Product (Samsca), whether or not it is considered causally related to the Medicinal Product.
Safety Information (Special Situations) | 90 days from the initiation of tolvaptan treatment
  Situations related to the use of an Otsuka product which may or may not be associated with an adverse event:
  * Maternal (pregnancy and breastfeeding) or paternal (via semen) exposure;
  * Exposure during breastfeeding;
  * Overdose/Incorrect dosage, misuse, abuse (e.g. patient sharing products);
  * Medication errors (e.g. patient took wrong dose);
  * Lack of therapeutic efficacy (e.g. the product doesn't work);
  * Occupational exposure (e.g.: nurse administering the product is exposed);
  * Cases of suspected transmission of infectious agents;
  * Use of suspected or confirmed falsified product(s) or quality defect of the product(s);
  * Withdrawal reactions;
  * Accidental exposure (e.g.: child takes parent's product);
  * Drug-drug/drug-food interactions;
  * Unintentional use of product in a non-approved population (e.g.: pediatric or geriatric population);
  * Disease progression/exacerbation of existing disease
Safety Information (Number of off-Label Use) | 90 days from the initiation of tolvaptan treatment
  Collecting any type of off-Label Use that refers to situations where a product is intentionally used for a medical purpose not in accordance with the authorized product information. Off-label use also includes the intentional use in non-authorized population categories not indicated in the label.
Safety Information (Serious Adverse Event) | 90 days from the initiation of tolvaptan treatment
  Any adverse drug experience/event occurring at any dose which
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or prolonged of existing hospitalization
  * results in persistent or significant disability or incapacity
  * is a congenital anomaly/birth defect
  * is medically significant.
Safety Information (Non-serious Adverse Events) | 90 days from the initiation of tolvaptan treatment
  All Adverse Events that do not meet the definition of a serious Adverse Event are considered non-serious Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Fukuta, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Pharmacovigilance Department, Osaka, Osaka, Japan